CLINICAL TRIAL: NCT01770756
Title: Improving the Willpower-based Self-care for Hypertension
Brief Title: FSU Hypertension Self-Care Training Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB terminated study
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSU-2012.8601
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2015-07

CONDITIONS: Hypertension
Keywords: Hypertension; High blood pressure; Willpower; Self care
MeSH Terms: conditions — Hypertension; Self-Control

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhancing willpower using active skills (Experimental): This group will use active tasks such as learning skills using hands to enhance willpower.
  Interventions: Behavioral: Self-Care Training
- Enhancing willpower using passive tasks (Experimental): This group will use passive tasks such as taking still postures to enhance willpower.
  Interventions: Behavioral: Self-Care Training

INTERVENTIONS:
Behavioral: Self-Care Training

SUMMARY:
The purpose of this study is to compare the effectiveness of two forms of self-care training on the overall health of adults with hypertension.

DETAILED DESCRIPTION:
The FSU College of Social Work and the Department of Psychology are seeking adults age 25 and older with a clinical diagnosis of hypertension for a randomized trial using willpower to manage high blood pressure. Voluntary participants will complete three phases: baseline, intervention, and post-treatment. Baseline phase includes a preliminary phone screening, fasting blood draw, physiological test (measuring heart rate variability, chest compression, etc.), and a psychosocial inventory. Intervention phase includes 8 weeks of once weekly trainings (approximately one hour long) to be held on a weekday evening. Participants will be randomly assigned to one of the two willpower groups and will be asked to rehearse the willpower method at least once daily for 30 minutes during these 8 weeks. Post-treatment phase includes two follow-up booster sessions (at week 12 and week 16) for refreshing willpower techniques, a follow-up fasting blood draw, a physiological test, and a psychosocial inventory.

Participation is completely voluntary and confidential. Volunteers completing each of the phases will be compensated $100 for their time. If someone is interested in participating, they should call our office at 850-645-0247 or email fsuwillpower@gmail.com.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hypertension
* Age 25 or older

Exclusion Criteria:

* Pregnancy
* Participation in other clinical trials or drug/behavioral treatment
* Previously participated in any other clinical trials/training on health-related behavior (tai-chi, yoga, nutritional education, yoga class)
* Kidney disease
* Cancer/chemotherapy, advanced HIV/AIDS, severe liver disease
* Severe ischemic heart disease (unstable angina, hospitalization for heart attack, coronary revascularization)
* Congestive heart failure
* Severe inflammatory/rheumatologic disorders (severe arthritis)
* Severe mental health diagnosis such as schizophrenia or bi-polar disorder
* Occurrence of any neurological disorders such as stroke or dementia
* Addicted to any legal/illegal drugs or alcohol without at least 1 year of sobriety
* Any infectious conditions such as pneumonia, traumatic wound, or surgery that may cause inflammation in the past 14 days

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Effects of two forms of self-care training on overall health of adults with hypertension | 20 weeks from beginning of training sessions

CONTACTS AND LOCATIONS:
Overall Officials: Amy L Ai, PhD, Principal Investigator — Florida State University
Locations (1):
- FSU College of Social Work, Tallahassee, Florida, United States